CLINICAL TRIAL: NCT00114673
Title: A Multicenter Study to Validate Cosmetic Outcome Scales Used to Assess Irregular Skin Pigmentation and Wrinkling
Brief Title: A Study to Validate Cosmetic Outcome Scales Used to Rate Uneven Skin Color and Wrinkling
Status: Completed | Type: Observational
Sponsor: Graceway Pharmaceuticals, LLC (Industry)
Other Study IDs: 1521-R850
Record Dates: First submitted 2005-06-16; First posted 2005-06-17 (Estimated); Last update posted 2007-02-19 (Estimated); Status verified 2006-01

CONDITIONS: Skin Wrinkling
Keywords: Uneven skin color; Wrinkles; Wrinkles and uneven skin color in the area around the eyes

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Skin chronically exposed to the sun may become damaged and then develop wrinkles and/or uneven skin color. The purpose of this research study is to evaluate a newly developed scale (grading tool) that rates wrinkles and uneven skin color. This newly developed scale will be used in future topical drug studies to measure these changes in the skin.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age

Exclusion Criteria:

* Have any disease of the skin, condition, or cosmetics around the eyes that may cause difficulty with the skin assessment using the scale to rate wrinkles and uneven skin color

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Tania J Phillips, M.D., Principal Investigator — Boston University
Locations (1):
- Boston, Massachusetts, United States